CLINICAL TRIAL: NCT01320865
Title: Biomarkers in Pulmonary Arterial Hypertension Treated With Nilotinib
Status: Withdrawn | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kewal Asosingh, Ph.D, Associate Staff, The Cleveland Clinic
Other Study IDs: Novartis AMN-107
Record Dates: First submitted 2011-03-18; First posted 2011-03-23 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: PAH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with PAH treated with nilotinib

SUMMARY:
The investigators hypothesize that bone marrow progenitor cells are mobilized into the circulation in PAH, home to the lungs and differentiate into mast cells, which promote vascular remodeling and vasoconstriction through release of renin and chymase. As a corollary to this, the investigators hypothesize that anti cKit tyrosine kinase inhibitor (TKI), nilotinib, provides clinical benefit to patients through inhibition of mast cell progenitor proliferation, mobilization and differentiation. To test this, the investigators will determine if mast cell progenitors and mast cell biomarkers are related to nilotinib clinical response. This will be an ancillary study, part of a placebo-controlled, double-blind multi center clinical trial of nilotinib in pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

This study is a substudy and subjects must be enrolled in the main trial:

See Study Efficacy, Safety, Tolerability and Pharmacokinetics (PK) of Nilotinib (AMN107) in Pulmonary Arterial Hypertension (PAH) In clinical trials. (clinical Trial ID NCT01179737)

http://clinicaltrials.gov/ct2/show/NCT01179737?

Exclusion Criteria:

Subjects are not enrolled in the main study:

See Study Efficacy, Safety, Tolerability and Pharmacokinetics (PK) of Nilotinib (AMN107) in Pulmonary Arterial Hypertension (PAH) In clinical trials. (clinical Trial ID NCT01179737)

http://clinicaltrials.gov/ct2/show/NCT01179737?term=tasigna+and+pulmonary+hypertension&rank=1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with PAH that are enrolled in the Nilotinib clinical trial. http://clinicaltrials.gov/ct2/show/NCT01179737?term=tasigna+and+pulmonary+hypertension&rank=1
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Measuring circulating markers of Nilotinib affect | within one year of the end of the study
  We will measure markers of mast cell activation in blood and urine before and during treatment with nilotinib.

SECONDARY OUTCOMES:
Evaluate effect of Nilotinib on the activation of mast cells. | within one year of the end of the study
  We will measure markers of mast cell activation in blood and urine before and during treatment with nilotinib. We will also look at the proliferation of mast cell progenitors and correlate this to clinical markers used to monitor this disease.

CONTACTS AND LOCATIONS:
Overall Officials: Kewal Asosingh, Ph.D, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Patterson KC, Weissmann A, Ahmadi T, Farber HW. Imatinib mesylate in the treatment of refractory idiopathic pulmonary arterial hypertension. Ann Intern Med. 2006 Jul 18;145(2):152-3. doi: 10.7326/0003-4819-145-2-200607180-00020. No abstract available. PMID 16847299
- [Background] Schermuly RT, Dony E, Ghofrani HA, Pullamsetti S, Savai R, Roth M, Sydykov A, Lai YJ, Weissmann N, Seeger W, Grimminger F. Reversal of experimental pulmonary hypertension by PDGF inhibition. J Clin Invest. 2005 Oct;115(10):2811-21. doi: 10.1172/JCI24838. PMID 16200212
- [Background] Dentelli P, Rosso A, Balsamo A, Colmenares Benedetto S, Zeoli A, Pegoraro M, Camussi G, Pegoraro L, Brizzi MF. C-KIT, by interacting with the membrane-bound ligand, recruits endothelial progenitor cells to inflamed endothelium. Blood. 2007 May 15;109(10):4264-71. doi: 10.1182/blood-2006-06-029603. Epub 2007 Feb 8. PMID 17289809
- [Background] Heath D, Yacoub M. Lung mast cells in plexogenic pulmonary arteriopathy. J Clin Pathol. 1991 Dec;44(12):1003-6. doi: 10.1136/jcp.44.12.1003. PMID 1791199
- [Background] Hamada H, Terai M, Kimura H, Hirano K, Oana S, Niimi H. Increased expression of mast cell chymase in the lungs of patients with congenital heart disease associated with early pulmonary vascular disease. Am J Respir Crit Care Med. 1999 Oct;160(4):1303-8. doi: 10.1164/ajrccm.160.4.9810058. PMID 10508822
- See also: See Study: Efficacy, Safety, Tolerabilitiy and PK of AMN 107 in PAH — http://clinicaltrials.gov/ct2/show/NCT01179737?term=tasigna+and+pulmonary+hypertension&rank=1